CLINICAL TRIAL: NCT05391165
Title: Effect of Back School-based Intervention on Non-specific Low Back Pain in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Associate professor in health sciences, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6009
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): ntervention based on the Back School was carried out for 8 weeks with a frequency of two sessions per week, with a total of 16 sessions lasting 45 min.
  Interventions: Behavioral: Back school
- Control group (No Intervention): I declare that I will not change my lifestyle during the study process.

INTERVENTIONS:
Behavioral: Back school — Intervention was carried out for 8 weeks with a frequency of two sessions per week, with a total of 16 sessions lasting 45 min. Of all the sessions, 14 had a practical focus and the other two had a theoretical focus. In the practical part, strengthening and stretching exercises were performed. In the theoretical part, self-management and pain neuroscience education were performed.
  Arms: Experimental group

SUMMARY:
The study consists of a theoretical and practical intervention based on the Back School. This intervention will be carried out over 8 weeks with a frequency of two sessions per week, for a total of 16 sessions of 45 minutes duration. Of all the sessions, 14 had a practical focus (strength and stretching exercises) and the other two had a theoretical focus (self-management techniques and pain neuroscience education). In addition, they had an initial session and a session at the end of the of the intervention in which measurements of the different variables were taken (The Visual Analogue Scale; Roland morris disability questionnaire scoring; Short Form 36 Health Survey; Tampa Scale Of kinesiophobia).These variables will be measured on two occasions, at the beginning of the study and at the end of the intervention, an average of 2 months.

The clinical practice guidelines highlight the importance of neck pain prevention through exercise an education. There are previous studies of the effects of theoretical and practical programmes based on back school on the lumbar region but not on the cervical region. Therefore, the aim of this study is to investigate the effects of a BS-based intervention on low back pain and functionality as well as kinesiophobia and quality of life in adults. The hypothesis previously hypothesised that this BS-based intervention would have positive effects on pain, functionality, kinesiophobia and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age. With non-specific low back pain for at least three months, with pain intensity (30-70 on a VAS).

Exclusion Criteria:

* History of cancer, spine infection, rheumatologic diseases, history of spine fracture, history of trauma, red flag signs including unwanted weight loss (exceeding 10 percent of the total body weight) in the past six months and fever, history of psychological disease and history of spine surgery, radiculopathy, anatomical and congenital disturbance.
* Missing more than two Back School sessions.
* Not being able to attend the measurement sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Through study completion, an average of 2 months.
  The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score).
Roland Morris Disability Questionnaire Scoring | Through study completion, an average of 2 months.
  The Roland Morris Disability Questionnaire Scoring (RMQ) is a 24-item patient-reported outcome measure that inquires about pain-related disability resulting from LBP. Items are scored 0 if left blank or 1 if endorsed, for a total RMQ score ranging from 0 to 24; higher scores represent higher levels of pain-related disability.
Short-Form Health Survey-36 | Through study completion, an average of 2 months.
  Short-Form Health Survey (SF-36) was used to measure quality of life.The SF-36 explores people's physical and mental health. It consists of 36 items that assessed eight dimensions of health status: social function, physical function, emotional role, physical role, mental health, vitality, physical pain, and general health. Scores ranged from 0 (worst health status) to 100 (best health status).
Tampa Scale Of Kinesiophobia. | Through study completion, an average of 2 months.
  This scale measures kinesiophobia. The total scale score ranges from 11 to 44, where 11 means no kinesiophobia and 44 means severe kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Beone Sport center, Pontevedra, Spain

REFERENCES:
- [Derived] Hernandez-Lucas P, Leiros-Rodriguez R, Mota J, Garcia-Soidan JL. Effects of a back school-based intervention on non-specific low back pain in adults: a randomized controlled trial. BMC Complement Med Ther. 2023 Jul 10;23(1):229. doi: 10.1186/s12906-023-04061-1. PMID 37430269